CLINICAL TRIAL: NCT06782438
Title: Evaluation of an Artificial Intelligence Algorithm Reducing Noise on Fast Whole-body Bone Tomoscintigraphy Acquisitions Recorded by a 360 Degree Cadmium-Zinc-Tellurid Camera
Acronym: IATOS2
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Achraf BAHLOUL, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI241
Record Dates: First submitted 2025-01-07; First posted 2025-01-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Bone Scan

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: artificial intelligence algorithm — to apply an artificial intelligence algorithm to treat the imaging

SUMMARY:
Recently, artificial intelligence algorithms reducing noise by deep learning have been developed with application to SPECT and PET images.

Many studies have reported the possibility of reducing the recording time in bone scintigraphy by applying artificial intelligence algorithms reducing noise

DETAILED DESCRIPTION:
Only two studies compared images denoised by a Deep Learning algorithm to those denoised by conventional filters (Gaussian and median filters). The first study was conducted only on patients, without phantom analysis and without taking into account the size of the lesions. The second study included an analysis on phantom and patients, but with application to planar images rather than to SPECT images that are increasingly used today

The hypothesis of our study conducted on phantom and patients is that an artificial intelligence algorithm reducing noise could replace the conventional filters usually used in bone SPECT for the denoising of scintigraphic images.

ELIGIBILITY:
Inclusion Criteria:

Patients who had a whole-body thee dimensions bone scan for rheumatological or oncological indications.

Exclusion Criteria:

Patients opposed to the use of their data

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a whole-body thee dimensions bone scan for rheumatological or oncological indications and non opposed to th use of their data
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
To compare imaging treated by the intelligence artificial algorithm with imaging treated with the traditionnal filter artificial algorithm | one day
  Quantification value on imaging measured with intelligence artificial algorithm compared with quantification value measured with conventional filter

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear Medicine Department, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Bahloul A, Rajadhas F, Doyen M, Lamash Y, Roth N, Roch V, Marie PY, Imbert L. A deep-learning noise reduction algorithm outperforms the spatial filters previously required for bone SPECT on a high-speed whole-body 360 degrees CZT-camera. EJNMMI Res. 2025 Dec 31. doi: 10.1186/s13550-025-01344-1. Online ahead of print. PMID 41474536